CLINICAL TRIAL: NCT01389999
Title: Validation of the French Version of the Back Belief Questionnaire
Acronym: BBQ
Status: Terminated | Type: Observational
Why Stopped: difficult recruitment curve
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2010/AD-02; 2011-A00270-41 (Other: ANSM)
Record Dates: First submitted 2011-07-07; First posted 2011-07-08 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Back Pain Lower Back Chronic
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic back pain patients: Patients who have had back pain for at least three months.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Each patient is asked to fill out several questionnaires: a french version of the BBQ, as well as the FABQ, the TAMPA score, and the Québec questionnaire, the Dallas score, the HAD score and a visual analog scale for pain.

SUMMARY:
The goal of this study is to carry out a transcultural validation of the Back Belief Questionnaire in order to assess its appropriateness for French-speaking populations.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has had back pain for at least 3 months

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting for back pain, present for at least three months.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08-29 (Actual); Study Completion 2014-08-29 (Actual)

PRIMARY OUTCOMES:
Change in French BBQ questionnaire score | after physical theraphy (3 months)
  The change in the BBQ score subsequent to physical therapy will be evaluated.

SECONDARY OUTCOMES:
Change in FABQ score | post physical therapy (3 months)
  The change in the FABQ questionnaire score following physical therapy will be evaluated.
Change in TAMPA score | post physical therapy (3 months)
  The change in the TAMPA score following physical therapy will be evaluated.
Change in Québec questionnaire score | post physical therapy (3 months)
  The change in the Québec questionnaire score following physical therapy will be evaluated.
Change in DALLAS questionnaire score | post physical therapy (3 months)
  The change in the DALLAS questionnaire score following physical therapy will be evaluated.
Change in HAD questionnaire score | post physical therapy (3 months)
  The change in the HAD questionnaire score following physical therapy will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, France

REFERENCES:
- [Result] Dupeyron A, Lanhers C, Bastide S, Alonso S, Toulotte M, Jourdan C, Coudeyre E. The Back Belief Questionnaire is efficient to assess false beliefs and related fear in low back pain populations: A transcultural adaptation and validation study. PLoS One. 2017 Dec 6;12(12):e0186753. doi: 10.1371/journal.pone.0186753. eCollection 2017. PMID 29211745